CLINICAL TRIAL: NCT07334990
Title: Impact of a Hypnotic Recording on Artifacts in 4D CT in the Context of Stereotactic Body Radiation Therapy for Lung Cancer
Acronym: HYPNOCT-4D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ET25-084
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stereotactic Body Radiation Therapy; Lung Lesions
Keywords: Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypnotic record (Experimental)
  Interventions: Other: Hypnotic record

INTERVENTIONS:
Other: Hypnotic record — The hypnotic audio recording will be played through the room's speakers. The hypnotic recording is structured in three stages, with a 5-minute induction phase, a 5-minute working phase, and finally a 5-minute return phase.

SUMMARY:
This is a single-center prospective cohort study evaluating the impact of a simple audio recording hypnosis system on the occurrence of artifacts on 4D CT scans in patients requiring SBRT radiotherapy for lung lesions (peripheral or central).

The primary objective of the study is to evaluate the use of a hypnotic recording on the reduction of artifacts in 4D CT scans for patients undergoing stereotactic body radiation therapy for lung cancer.

The secondary objectives are to evaluate:

* the impact of hypnotic recording on the reduction of artifacts on intrathoracic structures (trachea, main bronchi, diaphragm, lesions, heart, and lungs),
* the regularity of respiratory amplitude,
* the regularity of respiratory rate,
* the volume of Internal Target Volume (ITV),
* the reproducibility of ITV volume,
* patient satisfaction.

  1. Before this dosimetric scan, the patient will complete a self-administered questionnaire on anxiety: the HADS-A questionnaire (Hospital Anxiety and Depression Scale-only questions relating to anxiety).

     During this examination, the MERM explains the dosimetric scan procedure to the patient. After the immobilization system has been set up in accordance with the department's standard protocol, a 4D CT scan will be performed while asking the patient to breathe regularly. In the event of an artifact at the level of the lesion, a second 4D CT scan will be performed under the same conditions.
  2. The hypnotic audio recording will be played through the room's speakers. The hypnotic recording is structured in three stages, with a 5-minute induction phase, a 5-minute working phase, and finally a 5-minute return phase.

     After 5 minutes of playback, the 4D CT scan for the study is performed using the same acquisition parameters as the free 4D CT scan.
  3. Following the first radiotherapy session and for all patients included in the study, a 4D dosimetric scan will be performed using the hypnotic recording again, as described above, in order to assess the inter-fraction reproducibility of the ITV volume.

Following this second 4D CT scan under hypnosis, patient satisfaction will be assessed (using a Likert scale questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years,
* Indication for lung SBRT, peripheral or central lesion,
* Patient new to hypnosis (medical or stage hypnosis),
* Patient covered by social security or equivalent,
* Dated and signed consent form.

Exclusion Criteria:

* Indication for treatment with abdominal compression,
* Patient undergoing treatment for multiple lesions in the same treatment sequence,
* Patient with an ultra-central lesion (distance to the mediastinum < 2 cm),
* Patient already included in this protocol,
* Cognitive or physical disorders preventing the trial from proceeding smoothly,
* Patient with one or more active psychotic disorders (such as schizophrenia),
* Patients suffering from severe dissociative disorders,
* Patient who does not understand French or is deaf,
* Pregnant or breastfeeding women,
* Patient under guardianship or curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference between the proportion of 4D CT scans acquired under normal conditions and showing at least 1 artifact at the level of the lesion and the proportion of 4D CT scans acquired under hypnosis and showing >= 1artifact at the level of the lesion | Throught study completion, an average of 1 month

SECONDARY OUTCOMES:
The proportion of 4D CT scans showing at least one artifact in lung volume for both acquisition conditions (with and without hypnotic recording) | Throught study completion, an average of 1 month
The difference between the minimum and maximum respiratory amplitude for the two acquisition conditions (with and without hypnotic recording); | Throught study completion, an average of 1 month
The difference between the minimum and maximum respiratory rate for the two acquisition conditions (with and without hypnotic recording); | Until the end of the study
The difference in ITV volume between the two acquisition conditions (with and without hypnotic recording) | Throught study completion, an average of 1 month
The difference in ITV size, in the craniocaudal axis, on 4D CT scans acquired under hypnotic recording | Throught study completion, an average of 1 month
The satisfaction questionnaire score (5-point Likert scales) following the second 4D CT scan under hypnosis. | Throught study completion, an average of 1 month